CLINICAL TRIAL: NCT06341062
Title: The Application of Contrast-enhanced Ultrasound in Acute Kidney Injury in Intensive Care Unit
Brief Title: The Application of Contrast-enhanced Ultrasound in Acute Kidney Injury in ICU
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Cui Ligang, Chief Physician, Peking University Third Hospital
Other Study IDs: M2024078
Record Dates: First submitted 2024-03-17; First posted 2024-04-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Intensive Care Unit; Acute Kidney Injury; Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients recovering before hospital discharge: Recovery is defined as a return to normal serum creatinine and urine volume or more than 50% improvement in serum creatinine and/or urine volume from baseline
- Patients not recovering before hospital discharge: Non-recovery is defined as no significant improvement or further increase in serum creatinine and/or urine volume, the need for dialysis, or death.
  Interventions: Other: Renal microcirculation quantitatively assessed by Contrast-enhanced ultrasound

INTERVENTIONS:
Other: Renal microcirculation quantitatively assessed by Contrast-enhanced ultrasound — Renal microcirculation quantitatively assessed by Contrast-enhanced ultrasound before hospital discharge
  Groups: Patients not recovering before hospital discharge

SUMMARY:
The goal of this study is to quantitatively assess renal microcirculation changes by contrast-enhanced ultrasound and to obtain systemic hemodynamic information by ultrasound Doppler at the same time, to analyze the relationship between renal microcirculation changes and systemic hemodynamic changes, and to explore its predictive value in renal function recovery in patients with critical acute kidney injury. The main questions it aims to answer are:

1. To explore the quantitative parameters of contrast-enhanced ultrasound which can reflect the changes of renal microcirculation.
2. To explore the relationship between renal microcirculation and systemic hemodynamics.
3. To explore the value of renal microflow changes quantitatively evaluated by contrast-enhanced ultrasound in predicting renal function recovery.

DETAILED DESCRIPTION:
Quantitative analysis of cortical perfusion by contrast-enhanced ultrasound； Echocardiography； Quantitative results of renal artery and vein spectrum

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old;
* AKI was diagnosed < 24 hours after first admission to intensive care unit (ICU) and the expected length of stay in ICU ≥48 hours;
* Meet Kidney Disease Improving Global Outcomes (KDIGO) 2012 diagnostic criteria for acute kidney injury;
* Contrast-enhanced ultrasound was performed within 24 hours after diagnosis of acute kidney injury (AKI).

Exclusion Criteria:

* Known severe chronic kidney disease (CKD≥ stage 4) or undergoing hemodialysis treatment;
* Kidney transplantation or renal malignancy;
* Terminal stage of malignant tumor;
* Pregnancy;
* Renal artery stenosis or renal vein thrombosis;
* Allergy to contrast agent SonoVue(BraccoSpA, Milan, Italy) or its components, or the presence of severe cardiopulmonary insufficiency (e.g., right-to-left shunt heart disease or pulmonary systolic blood pressure >90mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Published contrast-enhanced ultrasound data from critically ill patients are limited. Through literature review, the area under the curve of contrast-enhanced ultrasound to predict kidney recovery in critically ill AKI patients is 0.72, and the width of confidence interval is 0.35. When α=0.05, the sample size N=34 is obtained by using PASS software. Considering the 20% shedding rate, 44 patients are expected to be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine values and/or urine output | Through study completion, an average of 7 days
  Complete recovery (defined as a return to normal serum creatinine and urine volume) and reversal of acute kidney injury (AKI) (more than 50% improvement in serum creatinine and/or urine volume from baseline), non-recovery included persistent AKI(no significant improvement or further increase in serum creatinine and/or urine volume, the need for dialysis, or death.)

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Cui, Dr, Principal Investigator — Department of Ultrasound, Peking University Third Hospital
Locations (1):
- Department of Ultrasound Diagnosis, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No